CLINICAL TRIAL: NCT04864288
Title: Value of Penile Elastography in Diagnosis of Patients With Erectile Dysfunction and Non-responders to Intra-corporal Injection
Status: Completed | Type: Observational
Sponsor: Ramzy Raafat Mohamed Mohamed Elnabarawy, MD, MSc, MRCS (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Ramzy Raafat Mohamed Mohamed Elnabarawy, MD, MSc, MRCS, Ramzy Elnabarawy, Cairo University
Organization: Cairo University (Other)
Other Study IDs: MS-182-2019
Record Dates: First submitted 2021-04-24; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: To Investigate the Value of Penile Elastography in the Diagnosis of Fibrosis of CC

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: male patients (age ≥ 21) with erectile dysfunction (ED) and non-responders to intracorporal injection
  Interventions: Device: Shear Wave Elastography
- 2: age matched thirty men with normal erectile function
  Interventions: Device: Shear Wave Elastography

INTERVENTIONS:
Device: Shear Wave Elastography — is a quantitative method in which the probe generates acoustic impulses through the tissue to create molecular vibration. These vibrations create shear waves so that elasticity might be calculated, because it is proportional to the speed of the waves

SUMMARY:
Penile erection is a neurovascular response that induces penile arterial dilatation, increased blood flow, and cavernous smooth muscles (CSM) relaxation; the enlarging corpora cavernosa compress the subtunical veins, against a rigid tunica albuginea, and entrap blood within the penis. Impaired CSM function can result in corporo veno-occlusive dysfunction (CVOD) and erectile dysfunction. Nevertheless, diagnostic tests, which can evaluate the status of CSM, are not clinically applicable. Penile elastography is a new promising tool that can assess the stiffness of the corpora cavernosa. Accordingly penile elastography can assess the status of the cavernous tissue and can distinguish patient with corporal fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* For group 1: Patients (age ≥ 21) have established sexual relationship for at least 3 months. These patients are complaining of ED and not responding to intracorporal injections (ICI).
* For group 2: Men (age ≥ 21) have an established sexual relationship for at least 3 months. These men have normal erectile function.

Exclusion Criteria:

* Peyronnie's disease, post-priapism corporal fibrosis, and clinically detected post traumatic corporal fibrosis, previous ICI therapy, history of penile and/or urethral surgery, liver cell failure, renal failure, heart failure, endocrinal diseases (e.g. thyroid- Adrenal), medications that may cause ED, and neurologic and psychotic disorders.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attendng Andrology clinic/ department and ultrasound unit at the radiology department at faculty of Medicine, Cairo University.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-09-28 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Penile elastography measurement data | 4 months
  Measurements in kPa to detect quantity of elastic tissue compared to fibrous tissue

CONTACTS AND LOCATIONS:
Overall Officials: Ramzy RM Elnabarawy, Principal Investigator — Kasr Alainy
Locations (1):
- Kasr Alainy outpatient clinics, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
To be made available upon request.

REFERENCES:
- [Background] Hassanin AM, Abdel-Hamid AZ. Cavernous smooth muscles: innovative potential therapies are promising for an unrevealed clinical diagnosis. Int Urol Nephrol. 2020 Feb;52(2):205-217. doi: 10.1007/s11255-019-02309-9. Epub 2019 Oct 15. PMID 31617065
- [Result] Dean RC, Lue TF. Physiology of penile erection and pathophysiology of erectile dysfunction. Urol Clin North Am. 2005 Nov;32(4):379-95, v. doi: 10.1016/j.ucl.2005.08.007. PMID 16291031
- [Result] Hamidi N, Altinbas NK, Gokce MI, Suer E, Yagci C, Baltaci S, Turkolmez K. Preliminary results of a new tool to evaluate cavernous body fibrosis following radical prostatectomy: penile elastography. Andrology. 2017 Sep;5(5):999-1006. doi: 10.1111/andr.12408. Epub 2017 Aug 8. PMID 28787549